CLINICAL TRIAL: NCT00310505
Title: Randomised Double Blind Dose Ranging Study of Amphotericin B in Visceral Leishmaniasis
Brief Title: Amphotericin B Treatment in Visceral Leishmaniasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS01MZP03
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Visceral Leishmaniasis
Keywords: visceral leishmaniasis; amphotericin B; Kala-azar
MeSH Terms: conditions — Leishmaniasis, Visceral

INTERVENTIONS:
Drug: Amphotericin B deoxycholate given as daily administration

SUMMARY:
This study is being conducted to assess the safety and efficacy of amphotericin B deoxycholate in doses of 0.75 mg/kg or 1.0 mg/kg for 15 doses. In each arm the drug is given in the conventional way every alternate day against the daily administration regimen being tested.

DETAILED DESCRIPTION:
This study is being conducted to assess the safety and efficacy of amphotericin B deoxycholate in doses of 0.75 mg/kg or 1.0 mg/kg for 15 doses. In each arm the drug is given in the conventional way every alternate day against the daily administration regimen being tested.

ELIGIBILITY:
Inclusion Criteria:

* Parasitologically proved kala-azar

Exclusion Criteria:

* HIV positive serology

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2003-01

PRIMARY OUTCOMES:
Final cure rate at six months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Kala-azar Medical Research Center, Muzaffarpur, Bihar, India

REFERENCES:
- [Derived] Sundar S, Chakravarty J, Rai VK, Agrawal N, Singh SP, Chauhan V, Murray HW. Amphotericin B treatment for Indian visceral leishmaniasis: response to 15 daily versus alternate-day infusions. Clin Infect Dis. 2007 Sep 1;45(5):556-61. doi: 10.1086/520665. Epub 2007 Jul 23. PMID 17682988